CLINICAL TRIAL: NCT03153696
Title: Application of Theory and Evidence to Promote Full Recovery From Pediatric Injury
Brief Title: Initial Evaluation of the Cellie Coping Kit for Children With Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meghan Marsac (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor-Investigator, Meghan Marsac, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-0187-P1G
Record Dates: First submitted 2017-05-02; First posted 2017-05-15 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cellie Intervention (Experimental): The Cellie Coping Kit intervention is grounded in empirical evidence regarding injury recovery. By utilizing parents as coaches, the Cellie Coping intervention can be initiated in the hospital and continued as the child recovers at home. The intervention's portable, engaging design and active partnership with parents as consistently available coaches, allows families to use the intervention anywhere (i.e., home, hospital, during procedures) ensuring the child is supported at the time the injury-related stressor arises. The Cellie Coping Intervention consists of 1) a stuffed toy to promote engagement, 2) caregiver book, and 3) coping cards. Skills are presented in a way usable by most parents and children without medical team support. In this condition, children and parents will be introduced to the Cellie Intervention immediately following the completion of the T1 measures.
  Interventions: Behavioral: Cellie Coping Kit Intervention
- Cellie Wait-list Control (Other): The Cellie Coping Kit intervention is grounded in empirical evidence regarding injury recovery. By utilizing parents as coaches, the Cellie Coping intervention can be initiated in the hospital and continued as the child recovers at home. The intervention's portable, engaging design and active partnership with parents as consistently available coaches, allows families to use the intervention anywhere (i.e., home, hospital, during procedures) ensuring the child is supported at the time the injury-related stressor arises. The Cellie Coping Intervention consists of 1) a stuffed toy to promote engagement, 2) caregiver book, and 3) coping cards. Skills are presented in a way usable by most parents and children without medical team support. In this condition, children and parents will be introduced to the Cellie Intervention via phone and mail following the completion of the T3 measures.
  Interventions: Behavioral: Cellie Coping Kit Intervention

INTERVENTIONS:
Behavioral: Cellie Coping Kit Intervention — The Cellie Coping Kit intervention is grounded in empirical evidence regarding injury recovery. By utilizing parents as coaches, the Cellie Coping intervention can be initiated in the hospital and continued as the child recovers at home. The intervention's portable, engaging design and active partnership with parents as consistently available coaches, allows families to use the intervention anywhere (i.e., home, hospital, during procedures) ensuring the child is supported at the time the injury-related stressor arises. The Cellie Coping Intervention consists of 1) a stuffed toy to promote engagement, 2) caregiver book, and 3) coping cards. Skills are presented in a way usable by most parents and children without medical team support.

SUMMARY:
The purpose of this study is to assess the feasibility (fidelity, acceptability, implementation, cost) of the Cellie Coping Kit for Children with Injury as well as to determine the intervention's efficacy (mechanisms of action and health outcomes).

DETAILED DESCRIPTION:
The goal of this study is to assess the Cellie Coping Kit for Injury intervention feasibility and initial efficacy.

Aim 1: Intervention Feasibility Assess intervention feasibility (implementation, cost, fidelity).

Aim 2: Intervention Efficacy (Mechanisms of Action and Health Outcomes): Conduct initial efficacy evaluation of the Cellie Intervention on mechanisms of action (adherence and coping behaviors) and health outcomes (physical recovery, HRQOL, emotional health).

Hypotheses: At 6-week follow-up (T2), compared to a Treatment as Usual (TAU) control group, parents in the intervention group will report greater adherence to medical discharge instructions (H2.1) and encourage their child to use a higher number of adaptive coping strategies (cognitive, active, support seeking; H2.2); children in the intervention group will generate a greater number of adaptive coping strategies (H2.3).

Hypotheses: At a 12-week follow-up (T3), compared to TAU, children in the intervention group will report better HRQOL and emotional health (H2.4); parents in the intervention group will report better child HRQOL and child emotional health (H2.5). Objective injury recovery scores will be higher for the intervention group (H2.6).

Method: 80 children with injury and one parent per child will participate in a pilot RCT with a wait-list control design. Participants will complete baseline assessments of targeted study variables prior to randomization (40 to the intervention; 40 to usual care) and then repeat measures 6 (T2), 12 (T3), and 18 weeks (T4) later. Those in the immediate intervention condition will initiate the intervention following the T1 assessment. Those in the wait-list condition will initiate the intervention following the T3 assessment.

ELIGIBILITY:
Inclusion Criteria:

* child has incurred an injury within the last month requiring medical attention
* one caregiver per child willing to participate
* sufficient English language skills to understand intervention and assessment materials
* access to internet or telephone for follow-up assessments

Exclusion Criteria:

* injury resulting from family violence

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Cellie Coping Kit Intervention | 6 weeks
  Feasibility will be primarily assessed via a self-report satisfaction score.

SECONDARY OUTCOMES:
Initial assessment of efficacy of Cellie Intervention on adherence | 6 weeks
  Compare intervention to wait-list control group on adherence
Initial assessment of efficacy of Cellie Intervention on coping behaviors | 6 weeks
  Compare intervention to wait-list control group on coping behaviors
Initial assessment of efficacy of Cellie Intervention on physical recovery | 12 weeks
  Compare intervention to wait-list control group on physical recovery
Initial assessment of efficacy of Cellie Intervention on HRQOL | 12 weeks
  Compare intervention to wait-list control group on HRQOL
Initial assessment of efficacy of Cellie Intervention on emotional health | 12 weeks
  Compare intervention to wait-list control group on emotional health

OTHER OUTCOMES:
Examine intervention timing effects | 18 weeks
  Examine differences in 12 week and 18 week outcomes on mechanisms of action and targeted health outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Marsac, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marsac ML, Sprang G, Guller L, Kohser KL, Draus JM Jr, Kassam-Adams N. A parent-led intervention to promote recovery following pediatric injury: study protocol for a randomized controlled trial. Trials. 2019 Feb 18;20(1):137. doi: 10.1186/s13063-019-3207-9. PMID 30777113